CLINICAL TRIAL: NCT06537518
Title: Adductor Canal Block With Dexamethasone Versus Adductor Canal Block With Systemic Dexamethasone in Arthroscopic Anterior Cruciate Ligament Repair
Brief Title: The Difference Between Using Local and General Dexamethasone in Arthroscopic Anterior Cruciate Ligament Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mahmoud Sharara, Lecturer of Anesthesiology, Pain, and ICU Department, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC 43-11-2023
Record Dates: First submitted 2024-07-26; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Calcium Dobesilate; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IV anesthetic Group (Active Comparator)
  Interventions: Drug: Dexamethasone injection; Drug: Bupivacaine 0.375% Injectable Solution
- Local anesthetic Group (Active Comparator)
  Interventions: Drug: Dexamethasone injection; Drug: Bupivacaine 0.5% Injectable Solution
- Control Group (Active Comparator)
  Interventions: Drug: Bupivacaine 0.375% Injectable Solution

INTERVENTIONS:
Drug: Dexamethasone injection — Dexamethasone, a potent glucocorticoid, decreases the inflammatory response, tissue damage, and pain after surgical procedures; which can be injected locally or Intravenously.
  Arms: IV anesthetic Group; Local anesthetic Group
Drug: Bupivacaine 0.375% Injectable Solution — Isobaric bupivacaine (0.375%) is injected into the adductor canal deeply to the sartorius muscle around the saphenous nerve after ensuring negative aspiration space.
  Arms: Control Group; IV anesthetic Group
Drug: Bupivacaine 0.5% Injectable Solution — 20 ml of Bupivacain 0.5% was mixed with dexamethasone 8 mg is injected into the adductor canal deeply to the sartorius muscle around the saphenous nerve after ensuring negative aspiration space.
  Arms: Local anesthetic Group

SUMMARY:
Arthroscopic knee injuries, such as the anterior cruciate ligament (ACL) injury, are common and often result in postoperative pain. Regional anesthetic techniques, such as femoral nerve block (FNB) and adductor canal block (ACB), can help alleviate pain and reduce opioid consumption. ACB, which blocks the saphenous nerve and obturator nerve branches, is preferred over FNB due to its potential to decrease mobility and increase falls risk. Dexamethasone, a potent glucocorticoid, is used as an adjuvant for ACB, but its perineural administration may carry neurotoxicity risks. Some pain physicians prefer intravenous administration to prolong the action of local anesthetics used in peripheral nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ACL injury;
* Patients in class I, II according to American Society of Anesthesiologists (ASA) classification.

Exclusion Criteria:

* Patients free of all Inclusion Criteria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reporting at least a 50% reduction in pain (measured by Numerical Rating Scale) post-arthroscopic ACL management. | 6 months
  Value of administration of dexamethasone enhancing the analgesic action of bupivacaine used in ACB after arthroscopic management of the ACL.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha faculty of Medicine, Banhā, El Qalyoubia, Egypt